CLINICAL TRIAL: NCT02329314
Title: The Evaluation of Glycyrrhizic Acid's Pesticide Effect in Treating Liver Damage (Retrospective Study）
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ShuGuang Hospital (Other)
Responsible Party: Principal Investigator, Chao Wu, postgraduate, ShuGuang Hospital
Other Study IDs: 2014-365-61-01
Record Dates: First submitted 2014-12-26; First posted 2014-12-31 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Liver Damage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Collect the details about hepatic dysfunctional patients induced by various etiology who have a usage of Glycyrrhizic Acid, then arrange and analyse the data to evaluate the clinical curative effect of glycyrrhizic acid.

DETAILED DESCRIPTION:
This experiment will screen and collect qualified cases from medical records in Shuguang Hospital.to collect the patients with liver injury in clinic, including (1) conforms to ALT>1.5 times the normal value or >70 IU/L, age 18 to 70 years of age, sex is not limited; (2) patients with viral hepatitis or cirrhosis of the liver, or autoimmune liver disease, or schistosomiasis, or drug-induced liver damage, or for other reasons clear or unclear leading to abnormal liver function ; (3) except for tumor patients. The index of liver function such as ALT, AST, Alb, et al are detected respectively before and after preventive treatment of the glycyrrhizic acid for liver injury ,and through the synthesizing of the single sample difference t test and clinical practice to analyze the clinical efficacy of glycyrrhizin intervention treatment of hepatic injury

ELIGIBILITY:
Inclusion Criteria:

1. conforms to ALT>1.5 times the normal value or >70IU/L, age 18 to 70 years of age, sex is not limited;
2. patients with viral hepatitis or cirrhosis of the liver, or autoimmune liver disease, or schistosomiasis, or drug-induced liver damage, or for other reasons clear or unclear leading to abnormal liver function ;

Exclusion Criteria:

1. patients with tumor;
2. pregnant or lactating women, and pregnancy may not take effective contraceptive measures;
3. complicated with serious heart, lung, gallbladder, kidney, endocrine, hematopoietic system and mental disease;
4. the researchers think that should not be selected for this test.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This experiment will screen and collect qualified casefrom medical records in Shuguang Hospital.to collect the patients with liver injury in clinic, including (1) conforms to ALT>1.5 times the normal value or >70IU/L, age 18 to 70 years of age, sex is not limited; (2) patients with viral hepatitis or cirrhosis of the liver, or autoimmune liver disease, or schistosomiasis, or drug-induced liver damage, or for other reasons clear or unclear leading to abnormal liver function ; (3) except for tumor patients.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Biochemical indexes measured before and after the interference | 1-4 weeks
  to measure biochemical indexes such as ALT, AST, ALB, TBiL, et al before and after the interference with Glycyrrhizic Acid

CONTACTS AND LOCATIONS:
Locations (1):
- Shuguang Hospital, Shanghai, Shanghai Municipality, China